CLINICAL TRIAL: NCT06990802
Title: Clinical and Cost-effectiveness of Learning Through Play Plus Culturally Adapted Cognitive Behaviour Therapy for Postnatal Depression in Nigeria
Acronym: LTP+CaCBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Coal City University, Nigeria (Unknown); Jos University Teaching Hospital, Nigeria (Unknown); Federal Medical Center, Abuja, Nigeria (Unknown)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Dr, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335g
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Postnatal Depression; Child Health
Keywords: Postnatal depression; Child health; Intervention; Parenting; Childbirth; Maternal mental health
MeSH Terms: conditions — Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP+CaCBT and TAU (Experimental): The LTP+CaCBT comprises 12 in-person sessions (90 minutes each) of intervention, which is the recommended duration for psychological interventions. LTP+CaCBT is manualised, and sessions will be delivered 'in-person' by non-specialist Community Health Workers (CHWs) in Nigeria. The CHWs will be trained to deliver the LTP+CaCBT under the supervision of Nigerian clinical psychologists and psychiatrists on a weekly basis. The proposed project adopts the World Health Organisation's (WHO) recommendations of task-shifting strategies to use non-specialists to tackle shortages of culturally knowledgeable mental health workforce in LMiCs, hence using CHWs.
  The experimental group will also receive Treatment As Usual (TAU). This includes participating services' regular treatment routine for postnatal depression. This is a standard patient care pathway, such as the service providers' routine assessment, management, and antidepressant prescriptions.
  Interventions: Behavioral: Learning Through Play plus Culturally adapted Cognitive Behaviour Therapy (LTP+CaCBT); Drug: Treatment as Usual (TAU)
- TAU alone (Active Comparator): Treatment As Usual (TAU) alone group will receive the participating services' regular treatment routine for postnatal depression. This is a standard patient care pathway, such as the service providers' routine assessment, management, and antidepressant prescriptions which is entirely different from LTP+CaCBT.
  Interventions: Drug: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Learning Through Play plus Culturally adapted Cognitive Behaviour Therapy (LTP+CaCBT) — LTP+CaCBT has two components. LTP is underpinned by Piaget's theory of cognitive development and Bowlby's theory of attachment. The CBT component uses active listening techniques, changing negative thinking, and guided discovery (i.e., Socratic questioning style to gently probe for cultural beliefs on mental health and stimulate alternative positive thinking). This includes a culturally adapted pictorial calendar devised for women, depicting successive stages of child well-being from 0-3 years, with illustrations of mother-child play and other culturally relevant activities that promote healthy parenting and mother-child attachment.
  Arms: LTP+CaCBT and TAU
Drug: Treatment as Usual (TAU) — TAU is the routine care currently available for the treatment of postnatal depression at the health care sites of intervention (e.g. diagnosis, management, antidepressant prescription and/or other forms of mental health care).

SUMMARY:
Background: We aim to examine the effectiveness of Learning Through Play and Cognitive Behaviour Therapy (LTP+CaCBT), a culturally appropriate psychosocial intervention to address postnatal depression among Nigerian women and improve the well-being of their children. Women of reproductive age (ages 16 to 49) comprise about 60 million of Nigeria's 230 million people. About 30% of these mothers experience postnatal depression. The global health challenge our research addresses is that one in three women worldwide experience postnatal depression and suicidal thoughts after childbirth, with long-term negative consequences on their children and families. Since 30% of Nigerian mothers suffer from postnatal depression, they have significant risks of transferring intergenerational mental health problems to their children. Over 250 million children are at risk of lacking developmental support in low- or middle-income countries, including Nigeria, due to postnatal depression, and this limits the children from reaching their full potential in life. The treatment gap for postnatal depression in Nigeria is huge due to a shortage of mental health specialists. Culturally appropriate, nonspecialist-delivered interventions are very limited in Nigeria. Our proposal aims to address this gap in treating postnatal depression using non-specialists called Indigenous Community Health Workers (CHWs), who are more culturally knowledgeable, as the World Health Organisation recommended in their task-shifting strategy.

Methods: We will evaluate the treatment, costs and implementation outcomes of LTP+CaCBT with 432 depressed mothers. Eligible participants (mother-child pairs) will be randomly selected to receive LTP+CaCBT and Treatment As Usual (TAU) or TAU alone. Our LTP+CaCBT intervention is a manualised 12-session (90-minute each) of mother-child play activities delivered in-person by CHWs under the supervision of clinical psychologists/psychiatrists. The eligible mothers (aged 16-49 years who have children between ages 0-36 months) will be assessed for depression before the intervention and then again at 4 months and 6 months afterwards. We will conduct interviews and focus group discussions to understand participants' and CHWs' experiences of the intervention

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* A mother with a child (0-3 years)
* Able to provide full consent for their participation
* A resident of the trial catchment areas
* Able to complete a baseline assessment
* Score 5 or above on Patient Health Questionnaire (PHQ-9)
* available for follow-up at 4 and 6 months post-enrolment

Exclusion Criteria:

* Less than 18 years
* Medical disorder that would prevent participation in a clinical trial, such as Tuberculosis or heart failure
* Temporary residents are unlikely to be available for follow-up
* Active suicidal ideation or any other severe mental disorder
* Patients currently undergoing severe mental health treatment
* Non-residents of the trial environs
* Unable to consent
* Unable to speak and understand English language
* Other significant physical or learning disability

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants - mothers of children between the ages of 0 and 3 years suffering from postnatal depression as a result of childbirth and parenting.
Enrollment: 432 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in postnatal depression is being assessed | Change is being assessed from baseline, end of intervention at 4 and at 6 months post-intervention
  Primary outcome measure would be assessed using the Patient Health Questionnaire (PHQ-9)

SECONDARY OUTCOMES:
Change in postnatal anxiety is being assessed | Change is being assessed from baseline, end of intervention at 4 and at 6 months post-intervention
  Secondary outcome measure would be assessed using the Generalised Anxiety Disorder (GAD7) scale
Change in health-related quality of life is being assessed | Change is being assessed from baseline, end of intervention at 4 and at 6 months post-intervention
  Outcome measure would be assessed using the Health-related Quality of Life scale (EuroQoL-5 Dimensions)
Change in social support is being assessed | Change is being assessed from baseline, end of intervention at 4 and 6 months post-intervention
  Outcome measures would be assessed using the Oslo Social Support Scale
Change in service satisfaction is being assessed | Change is being assessed from baseline, end of intervention at 4 and 6 months post-intervention
  Outcome measure would be assessed using the brief Verona Service Satisfaction Scale
Change in child physio-emotional development is being assessed | Change is being assessed from baseline, end of intervention at 4 and 6 months post-intervention
  Outcome measure would be assessed using the Ages and Stages Social-Emotional Questionnaire
Change in mother-child attachedment is being assessed | Change is being assessed from baseline, end of intervention at 4 and 6 months post-intervention
  Outcome measures would be assessed using the Maternal Attachment Inventory
Change in service satisfaction is being assessed | Change is being assessed at end of intervention at 4 months post-intervention
  Outcome measure would be assessed using the brief Verona Service Satisfaction Scale

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.